CLINICAL TRIAL: NCT01750502
Title: MIF Gene Polymorphism in Coronary Heart Disease：Clinical Meaning
Brief Title: The Clinical Diagnosis Meaning of MIF in Coronary Heart Disease
Status: Completed | Type: Observational
Sponsor: Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, JiFei Tang, Director, Wenzhou Medical University
Other Study IDs: wenzhouhp
Record Dates: First submitted 2012-11-24; First posted 2012-12-17 (Estimated); Results first posted 2015-03-04 (Estimated); Last update posted 2015-03-04 (Estimated); Status verified 2015-02

CONDITIONS: Coronary Heart Disease
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The biospecimen is blood that taken from cubital vein.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- coronary-artery-disease group: Participants, who are diagnosed as coronary-artery-disease which including acute coronary syndromes and stable ischemic heart disease, will receive at least one stent.
- non-coronary-artery-disease group: Participants, who are diagnosed as non-coronary-artery-disease without acute coronary syndromes and stable ischemic heart disease, will not receive stent.

SUMMARY:
Macrophage migration inhibitory factor (MIF) is a pleiotropic cytokine that promote the inflammatory response.In animal studies, it has been found that MIF is released in the ischaemic heart, promoting glucose uptake and protecting the heart from ischaemia-reperfusion injury.The MIF concentration, influenced by age and myocardial ischemia, have different impact on myocardial functional recovery after ischemia.Therefore, the purpose of this experiment is to study the clinical significance of MIF in patients with coronary heart disease.

DETAILED DESCRIPTION:
MIF is a pleiotropic cytokine that promote the inflammatory response. MIF is expressed in several cell types,including monocytes/macrophages, vascular smooth muscle and cardiomyocytes, and is released on stimulation from pre-formed storage pools. A foreign study reported that MIF had demonstrated to offer protection from I/R-injury by activating adenosine monophosphate-activated protein kinase (AMPK) and inhibiting c-Jun Nterminal kinase (JNK)-induced apoptosis of cardiomyocytes. In addition, animal experiments showed that MIF was reduced in aged heart compared with young heart. Coronary heart disease is a chronic ischemic disease, in which MIF may play as a protective factor during the whole procedure.

We observed individuals who will be taking coronary angiography during the hospitalization. Individuals will be assigned to coronary-artery-disease group, which included acute coronary syndromes and stable ischemic heart disease, or non-coronary-artery-disease group, according to coronary angiography. All participants will be extracted 3ml blood sample 5 minutes before coronary angiography. Coronary-artery-disease group will be taken another two blood samples, 5 minutes after the opening of the balloon and 5 minutes after the stents have been implanted, respectively.

ELIGIBILITY:
Inclusion Criteria:

Control group:

1. enroll individuals who confirmed by coronary angiography without coronary heart
2. The age between 20 and 80 years old.
3. Alanine aminotransferase(ALT):10-55U/L, Aspartate aminotransferase(AST):0-60U/L
4. Glucose(GLU-S):3.9-6.1mmol/L
5. Triglycerides(TRIG):0.56-1.7mmol/L, cholesterol(CHOL):3.1-5.2mmol/L, High density lipoprotein(HDL):0.78-1.96mmol/L, High density lipoprotein(LDL):2.07-3.1mmol/L

Experimental group:

1. enroll individuals who confirmed by coronary angiography for coronary heart
2. The age between 20 and 80 years old.
3. ALT:10-55U/L,AST:0-60U/L
4. GLU-S:3.9-6.1mmol/L
5. TRIG:0.56-1.7mmol/L,CHOL:3.1-5.2mmol/L,HDL:0.78-1.96mmol/L,LDL:2.07-3.1mmol/L

Exclusion Criteria:

1. Inflammatory diseases,such as rheumatoid arthritis,sepsis,asthma and acute respiratory distress syndrome.
2. Diabetes

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Second Hispital of Wenzhou Medical College outpatient and inpatient
Sampling Method: Probability Sample
Enrollment: 256 (Actual)
Dates: Start 2012-05; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jifei Tang, MD, Principal Investigator — Wenzhou Medical University
Locations (1):
- Second Hispital of Wenzhou Medical College, Wenzhou, Zhejiang, China

REFERENCES:
- [Derived] Qian L, Wang XY, Thapa S, Tao LY, Wu SZ, Luo GJ, Wang LP, Wang JN, Wang J, Li J, Tang JF, Ji KT. Macrophage migration inhibitory factor promoter polymorphisms (-794 CATT5-8): Relationship with soluble MIF levels in coronary atherosclerotic disease subjects. BMC Cardiovasc Disord. 2017 Jun 2;17(1):144. doi: 10.1186/s12872-017-0570-x. PMID 28578664
- [Derived] Ji K, Wang X, Li J, Lu Q, Wang G, Xue Y, Zhang S, Qian L, Wu W, Zhu Y, Wang L, Liao L, Tang J. Macrophage migration inhibitory factor polymorphism is associated with susceptibility to inflammatory coronary heart disease. Biomed Res Int. 2015;2015:315174. doi: 10.1155/2015/315174. Epub 2015 Mar 4. PMID 25821795

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Sequencing was carried out after polymerase chain reaction with DNA specimens from 186 volunteers without CHD and 70 patients with CHD. CHD was confirmed by Coronary Angiography (CAG).
Period: Overall Study
Arm/Group | Coronary-artery-disease Group | Non-coronary-artery-disease Group
Started | 70 | 186
Completed | 70 | 186
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Coronary-artery-disease Group | Non-coronary-artery-disease Group | Total
Number analyzed (Participants) | 70 | 186 | 256
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 59 | 151 | 210
  >=65 years | 11 | 35 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.02 (8.57) | 65.9 (10.03) | 64.96 (9.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 97 | 130
  Male | 37 | 89 | 126
Region of Enrollment [Number; unit: participants]
  China | 70 | 186 | 256
Hypertension [Number; unit: participants]
  Hypertension | 46 | 111 | 157
  Not Hypertension | 24 | 75 | 99
HDL-C [Mean (Standard Deviation); unit: mmol/L] | 1.01 (0.23) | 0.98 (0.22) | 0.99 (0.22)
LDL-C [Mean (Standard Deviation); unit: mmol/L] | 2.47 (0.74) | 2.4 (1.43) | 2.44 (0.98)

OUTCOME MEASURES:

1. Primary Outcome: Comparison Between Coronary-artery-disease Group and Non-coronary-artery-disease Group on MIF Concentration
Description: Participants will be extracted 3ml blood before surgery 5 minutes,detection MIF concentration on two groups.We hypothesis that the experimental group will be higher than control group.
Time Frame: Before surgery 5 minutes
Population: All participants drawn from hospital inpatient cardiovascular medicine between June 2012-January 2013.This analysis was per protocol, but not intention to treat.Because the number of CHD group is less than the normal group during hospitalization.
Measure: Median (Standard Deviation); unit: MIF Concentration,ug/L
Arm/Group | Non-coronary-artery-disease Group | Coronary-artery-disease Group
Number analyzed (Participants) | 186 | 70
MIF Concentration,ug/L | 48.08 (6.48) | 66.79 (6.29)

2. Secondary Outcome: Comparison the Change of MIF Before and After Percutaneous Coronary Intervention （PCI） at the Patients Who Are Acute Coronary Syndromes and Stable Ischemic Heart Disease
Description: Percutaneous Coronary Intervention are extracted 3 times including before surgery 5 minutes , 5 minutes after the opening of the balloon and after surgery 5 minutes ,and detection MIF concentration .
Time Frame: 3 times including before surgery 5 minutes, 5 minutes after the opening of the balloon and after surgery 5 minutes
Population: Coronary-artery-disease Group does not include myocardial infarction, 21 patients were acute myocardial infarction participants.
Measure: Mean (Standard Deviation); unit: MIF Concentration , ug/L
Groups:
- Before Surgery 5 Minutes; After Surgery 5 Minutes: Participants, who are diagnosed as coronary-artery-disease with acute coronary syndromes or stable ischemic heart disease,they Were undergoing PCI.
- 5 Minutes After the Opening of the Balloon: Participants, who are diagnosed as coronary-artery-disease which including acute coronary syndromes and stable ischemic heart disease, will receive at least one stent.
Arm/Group | Before Surgery 5 Minutes | After Surgery 5 Minutes | 5 Minutes After the Opening of the Balloon
Number analyzed (Participants) | 21 | 21 | 21
MIF Concentration , ug/L | 85.51 (6.44) | 85.40 (7.18) | 84.7 (5.21)

3. Other Pre Specified Outcome: Comparison With MIF-173G/C Genotypes of CHD Patients and Controls.
Time Frame: Before surgery
Measure: Number; unit: participants
Arm/Group | Coronary-artery-disease Group | Non-coronary-artery-disease Group
Number analyzed (Participants) | 70 | 186
participants
  Genotypes of CC | 10 | 6
  Genotypes of CG | 14 | 44
  Genotypes of GG | 46 | 136

4. Other Pre Specified Outcome: Comparison of MIF-173G/C Alleles of CHD Patients and Controls.
Time Frame: Before surgery
Population: as for outcome 1
Measure: Number; unit: alleles
Arm/Group | Non-coronary-artery-disease Group | Coronary-artery-disease Group
Number analyzed (Participants) | 186 | 70
alleles
  alleles of G | 316 | 106
  alleles of C | 56 | 34

ADVERSE EVENTS:
Arm/Group | Coronary-artery-disease Group | Non-coronary-artery-disease Group
Serious Adverse Events (participants affected / at risk) | 0/70 | 0/186
Other Adverse Events (participants affected / at risk) | 0/70 | 0/186

LIMITATIONS AND CAVEATS:
There are some limitations to this research. First, the sample size was relative small. Second,no participants were retrospectively analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less